CLINICAL TRIAL: NCT00231829
Title: A Pilot Phase II Trial of Celecoxib in Patients With Grade 2 or 3 Endometrioid-type, Clear Cell, and Papillary Serous Uterine Cancers
Brief Title: A Pilot Study of Celecoxib in Patients With Grade 2 or 3 Uterine Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to reported toxicity of Celecoxib at high doses
Sponsor: Mark H. Einstein (Other)
Collaborators: Pharmacia (Industry)
Responsible Party: Sponsor-Investigator, Mark H. Einstein, Director, Clinical Research for Women's Health, Montefiore Medical Center
Organization: Montefiore Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MMC-03-04-084
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Uterine Cancer
Keywords: Treatment; Uterine Papillary Serous Carcinoma; Clear Cell Carcinoma; COX-2 Inhibitors
MeSH Terms: conditions — Uterine Neoplasms; Adenocarcinoma, Clear Cell | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
Expression of COX-II has been identified in many types of human cancers. Uterine cancer is the most common gynecologic cancer in the US and there has been an increase in uterine cancer deaths over the past decade mainly due to the difficulty in treating recurrences in the more aggressive histologic types. The study co-investigators have also identified COX-II expression in grade 2 and 3 endometrioid-type, clear cell, and papillary serous types of uterine cancers. Upregulation of COX-II may control the cell cycle by regulating the proliferative capacity of neoplastic endometrial cells. This is a Phase II pre-post intervention comparison study in eligible patients looking at the effects of a COX-II inhibitor on uterine cancer. The patients whose endometrial biopsy shows grade 2 or 3 endometrioid-type, clear cell, and papillary serous types of uterine cancers will be put on a selective COX-II inhibitor, Celebrex (Celecoxib) until the day of their surgery. We hypothesize that Celecoxib will downregulate the expression of COX-II in these tumor types as it does in other similar tumors. We also hypothesize that apoptosis, as measured with the TUNEL assay, will be increased in areas with less COX-II expression and should be inversely proportional to cellular p21 expression. We hypothesize COX-related gene expression will be altered thus suggesting an up- or down-regulation of these genes in the end-organ tissue. Documenting downregulation of COX-II enzyme and altered gene expression in endometrial carcinoma after treatment with Celecoxib may result in further prospective studies using selective COX-II inhibitors as effective, well-tolerated chemotherapeutic agents in these uterine cancers that are resistant to many current therapies.

DETAILED DESCRIPTION:
Endometrial cancer is the most common gynecologic cancer in the United States. The number of deaths from endometrial cancer has risen 128% since 1987. In 2001, an estimated 38,300 women will develop endometrial cancer (ACS Facts and Figures) and an estimated 6,600 women will die from endometrial cancer. Preinvasive and well-differentiated endometrial cancers are hormonally driven and often cured with surgery alone. Higher-grade tumors are usually not hormonally driven and proliferate via unknown mechanisms. These tumors are largely responsible for the rising death rate. Responses to toxic treatment protocols for recurrent endometrial cancer are dismal. Unfortunately, these post-menopausal women also often have comorbidities, which limit their eligibility for current chemotherapy and radiotherapy treatments.

Expression of COX-II has been identified in many human cancers including: colon cancer, gastric cancer, esophogeal cancer, bladder cancer, head and neck cancer, liver cancer, pancreatic cancer, prostate cancer and breast cancer. COX-II expression is also strongly expressed in the primary tumor and metastasic site in human cervical cancer. COX-II may influence cell cycle control by upregulating the proliferative capacity of neoplastic endometrial cells. Furthermore, COX-II inhibitors inhibit tumor proliferation even in cells that do not express COX. This suggests an alternative mechanism of action not yet defined that may play a role in inhibiting the growth of cancer tissue.

The enhanced expression of COX-II has led investigators to use COX-II inhibitors in the prevention and/or treatment of colon and prostate cancers both in vivo and in vitro. Celecoxib is now FDA approved for chemoprevention of colon cancer in familial adenomatous polyposis patients. If it can be shown that COX-II is downregulated by COX-II inhibitors in endometrial cancer, they may offer similar chemopreventative or chemotherapeutic potentials that have already been proven in colon cancer.

COX-II enzyme activity may not always correlate with end organ gene expression. Multiple genes have been implicated in apoptotic pathways and are affected by COX-II inhibitors. NS-398, a selective COX-II inhibitor causes elevations in APC expression and downregulation of c-myc. Prostate apoptosis response 4 (Par-4) levels are increased in cells treated with COX inhibitors. PTEN and hMLH1 are genes which are implicated in malignant transformation of endometrial tissue. 5-Lipooxygenase (5-LOX) is often correlated with COX-I and COX-II. Thus, in addition to COX-I and COX-II, these are good candidate genes to study the effects of COX-II inhibitors on uterine cancers.

Preliminary Data Since COX-II expression is seen in the endometrium and in other hormonally-dependent tumors, we have investigated the expression of COX-II in endometrial cancer. Our preliminary studies on 41 fixed samples of benign and neoplastic endometrium revealed that COX-II was not expressed in benign endometrial tissue, stains minimally (~1% of tumor cells) in well-differentiated endometrial carcinomas, and stains most strongly in poorly-differentiated carcinomas (~12% of tumor cells, most staining strongly). COX-II is expressed in all poorly differentiated uterine cancers. Our study also demonstrated that COX-II was also strongly expressed in uterine papillary serous carcinomas (UPSC) as well as clear cell carcinomas of the uterus. These findings were confirmed by Ferrandina, et al. A small percent of our patients as well as the patients in the Ferrandina study have only 1+ or 1-5% staining. These 'low-expressers' only made up 1/13 (7.7%) of our patients.

COX-II expression in endometrial carcinoma has a slight inverse correlation with apoptosis (r=-0.534). However, COX-II expression in endometrial carcinoma correlated with lymphovascular invasion (r=0.69) and depth of invasion (r=0.68). There was no correlation between COX-II expression and ER (r=0.03) or PR (r=-0.02). The presence of a poorly-differentiated tumor may imply a hormonally-independent pathway resulting in de-differentiation. In summary, our preliminary data reveals that COX-II expression is high in grade 2 and 3 endometrioid-type endometrial cancers, as well as UPSC and clear cell subtypes and is correlated with known clinical prognostic factors.

Expression of COX-II has been identified in many types of human cancers. Uterine cancer is the most common gynecologic cancer in the US and there has been an increase in uterine cancer deaths over the past decade mainly due to the difficulty in treating recurrences in the more aggressive histologic types. The study co-investigators have also identified COX-II expression in grade 2 and 3 endometrioid-type, clear cell, and papillary serous types of uterine cancers. Upregulation of COX-II may control the cell cycle by regulating the proliferative capacity of neoplastic endometrial cells. This is a Phase II pre-post intervention comparison study in eligible patients looking at the effects of a COX-II inhibitor on uterine cancer. The patients whose endometrial biopsy shows grade 2 or 3 endometrioid-type, clear cell, and papillary serous types of uterine cancers will be put on a selective COX-II inhibitor, Celebrex (Celecoxib) until the day of their surgery. The expression of COX-II and p21 will be quantified after treatment with Celecoxib in eligible patients. This expression will be evaluated by performing immunohistochemical staining on the endometrial biopsy (pre-intervention) and the hysterectomy specimen (post-intervention). Apoptosis, evaluated by the terminal deoxynucleotidyl transferase (TdT)-mediated dUTP- digoxigenin nick end-labeling (TUNEL) assay, will also be evaluated and compared to COX-II expression in endometrial cancer in the two specimens, endometrial biopsy (pre-intervention) and uterus (post-intervention). In addition to IHC analysis and apoptosis, gene expression of COX-related genes in the post-intervention uterine specimens will. This gene expression will be compared to matched controls who were not treated with a COX-II inhibitor. COX-II expression will be correlated with established clinical prognostic factors including lymphovascular invasion, depth of myometrial invasion and lymph node involvement. We hypothesize that Celecoxib will downregulate the expression of COX-II in these tumor types as it does in other similar tumors. We also hypothesize that apoptosis, as measured with the TUNEL assay, will be increased in areas with less COX-II expression and should be inversely proportional to cellular p21 expression. Additionally, COX-II inhibitors affect apoptotic pathways even in cells that do not express COX-II. For low expressing cells, COX-II inhibitor activity may be better documented with apoptosis. We hypothesize COX-related gene expression will be altered thus suggesting an up- or down-regulation of these genes in the end-organ tissue. Documenting downregulation of COX-II enzyme and altered gene expression in endometrial carcinoma after treatment with Celecoxib may result in further prospective studies using selective COX-II inhibitors as effective, well-tolerated chemotherapeutic agents in these uterine cancers that are resistant to many current therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* Histologically confirmed uterine cancer of the following histologic types: grade 2 or grade 3 endometrioid-type, clear cell, or papillary serous types. The pre-therapy samples come from either an endometrial sampling (e.g. pipelle) or dilation and curettage of the uterus with or without hysteroscopy. Unstained slides of the primary tumor, a primary tumor block, or cytologic preparation must be available for review. COX-II expression is seen in the majority of patients with these tumor types. Effects of COX-II inhibitors occur even in the absence of COX-II expression and will be measured with other IHC staining, apoptosis studies and gene expression. Therefore, patients will not be tested for COX-II expression preoperatively in order to include them in the study.
* Disease status: Only patients with clinical stage I or stage II disease will be eligible.
* Negative urine pregnancy test in women of child-bearing potential (within 14 days of the initiation of Celebrex).
* All eligible patients need to have a Zubrod/ECOG/GOG performance status ≤2 that permits surgery, with or without staging, as indicated.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Celecoxib is contraindicated in patients with known hypersensitivity to Celecoxib. Celecoxib should not be given to patients who have demonstrated allergic-type reactions to sulfonamides. Celecoxib should not be given to patients who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs.
* Concurrent therapy: Patients who have had daily usage of any form of NSAID or aspirin prior to endometrial biopsy will be excluded from this study.
* Selective COX-II inhibitors have some activity on the gastrointestinal mucosa. Although Celecoxib is not contraindicated in patients with peptic ulcer disease, these patients will be excluded to avoid any untoward gastrointestinal side effects.
* There is no information regarding the use of Celecoxib in patients with advanced renal disease. Therefore, treatment with Celecoxib is not recommended in these patients.
* Patient has impairment of hepatic, renal or hematologic function as defined by the following baseline laboratory values performed <= 4 weeks prior to the study:

  * Serum SGOT and/or SGPT > 2.5 times the institutional upper limit of normal (IULN).
  * Total serum bilirubin > 1.5 mg/dL.
  * History of chronic active hepatitis or cirrhosis.
  * Serum creatinine > 2.0 mg/dL.
  * Platelets < 100,000/mm3
  * Absolute neutrophil count (ANC) < 1500/mm3
  * Hemoglobin < 8.0 g/dL
  * PT/PTT within normal range
  * Pregnant or nursing women are excluded. Women of child-bearing potential must agree to use a chemical or barrier contraceptive during the dosing portion of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23
Dates: Start 2003-04; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
To compare COX-II expression in grade 2 or grade 3 uterine cancers treated with Celecoxib, following endometrial biopsy (pre-intervention) and after hysterectomy (post-intervention)

SECONDARY OUTCOMES:
o To confirm the safety and tolerability of Celecoxib in this patient population.
o To evaluate alterations in the cell cycle pre- and post-intervention with Celecoxib.
o To evaluate apoptosis pre- and post-intervention using the TUNEL method.
o To evaluate the relationship between COX-II expression, apoptosis, p21 with clinical prognostic factors.
o To evaluate COX-related gene expression in the post-intervention uterine tissue by RT-PCR and compare to untreated matched controls.

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Einstein, M.D., M.S., Principal Investigator — Montefiore Medical Center and Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Cao QJ, Einstein MH, Anderson PS, Runowicz CD, Balan R, Jones JG. Expression of COX-2, Ki-67, cyclin D1, and P21 in endometrial endometrioid carcinomas. Int J Gynecol Pathol. 2002 Apr;21(2):147-54. doi: 10.1097/00004347-200204000-00007. PMID 11917224